CLINICAL TRIAL: NCT05185011
Title: A Phase I Clinical Study of the Pharmacokinetics and Safety of TPN171H Tablets in Subjects With Mild Liver Insufficiency, Moderate Liver Insufficiency and Normal Liver Function
Brief Title: Study of the Pharmacokinetics and Safety of TPN171H Tablets in Subjects With Mild ,Moderate Hepatic Insufficiency and Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPN171H-09
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-12

CONDITIONS: Erectile Dysfunction; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Erectile Dysfunction; Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild hepatic impairment (Experimental): Subjects with mild hepatic impairment
  Interventions: Drug: TPN171H
- moderate hepatic impairment (Experimental): Subjects with mild moderate impairment
  Interventions: Drug: TPN171H
- healthy volunteers (Experimental): Subjects with normal hepatic function
  Interventions: Drug: TPN171H

INTERVENTIONS:
Drug: TPN171H — 10 mg TPN171H tablets，single dose

SUMMARY:
The study aims to investigate and compare the effect of TPN171H on subjects with mild and moderate hepatic impairment compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Hepatic Insufficiency Participants：

1. Signing the informed consent forms；
2. Take proper contraceptive during the study and within 6 months after the study completed;
3. 18 years to 65 years (inclusive)；
4. Male≥50kg，femal≥45kg, Body mass index should be between 18 and 30 kg/m2 (inclusive)；
5. No medication was used before screening，or stable medication for 4 weeks. Liver cirrhosis；
6. Child-Pugh class A or Child-Pugh class B, liver function impairment caused by previous primary liver disease (drug-induced liver injury was excluded)；
7. The clinical diagnosis was liver cirrhosis.

Normal liver function Participants：

1. Signing the informed consent forms；
2. Take proper contraceptive during the study and within 6 months after the study completed;
3. 18 years to 65 years (inclusive)；
4. Male≥50kg，femal≥45kg, Body mass index should be between 18 and 30 kg/m2 (inclusive)；
5. No medication was used before screening；
6. Clinical laboratory tests during the screening period were normal，or the abnormality has no clinical significance.

Exclusion Criteria:

1. Allergic constitution；
2. Patients who have a history of NAION, or with a known genetically degenerative retinopathy, including retinitis pigmentosa；
3. Patients with alcohol addiction or persistent abuse of drugs of dependence;
4. Smoking more than 5 cigarettes per day within 3 months prior to screening；
5. Drug abuse within 3 months prior to screening，or the long-term use of benzodiazepine medications；
6. Blood donation (or blood loss) ≥200mL, or receiving whole blood transfusions or erythrocyte suspension transfusions within 3 months prior to the screening；
7. Patients with severe or clinically significant infections, traumas, and major trauma surgery within 4 weeks before screening;
8. Participated in any other intervention clinical trial within 1 months before screening；
9. Within 28 days before screening, inhibitors or inducers of CYP3A4 were used；
10. have a scheduled surgical plan during the study period;
11. Patients with clinically significant ECG abnormalities；
12. Creatinine clearance <60ml/min;
13. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial；
14. Screening positive for viral hepatitis (including hepatitis B and C), HIV or syphilis (normal liver function only) ；
15. Urine drug screening positive；
16. Any factors that the investigator considers inappropriate for participation in the study；

    Additional exclusion criteria for subjects with hepatic insufficiency (those who meet any of the followings are ineligible):
17. History of liver transplant;
18. History of any serious diseases, other than primary liver diseases, or history of disorders and/or clinically significant abnormal laboratory findings that, as judged by the investigator, may affect the results of the study, including but not limited to the history of diseases in the circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases;
19. Subjects with liver failure, acute liver injury ,or subjects with cirrhosis complicated with hepatocellular carcinoma or symptomatic hepatic encephalopathy, etc., are deemed as unsuitable for this study by the investigator；
20. ALT or AST >10*ULN，NE#<0.75*10^9/L,HGB<60g/L，AFP >100ng/ml；
21. Positive for HIV antibody screening; a rapid plasma reagin (RPR) test is required for a subject who tests positive for syphilis antibodies, and the subject should be excluded if the RPR result is also positive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 72 hours after dosing
  Maximum Plasma Concentration (Cmax) will be compared between normal hepatic function patients and mild or moderate hepatic dysfunction patients
Area under the plasma concentration versus time curve from single dosing time extrapolated to infinity（AUC0-∞） | 72 hours after dosing
  Area under the plasma concentration versus time curve from single dosing time extrapolated to infinity（AUC0-∞） will be compared between normal hepatic function patients and mild or moderate hepatic dysfunction patients
Area under the plasma concentration versus time curve from the last time of dosing to the last measurable concentration （AUC0-t） | 72 hours after dosing
  Area under the plasma concentration versus time curve from the last time of dosing to the last measurable concentration （AUC0-t） will be compared between normal hepatic function patients and mild or moderate hepatic dysfunction patients

SECONDARY OUTCOMES:
Adverse events | From administration of study drug through 7 days after administration of study drug
  Number of Participants With Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Hua Ding, MD, Study Chair — The First Affiliated Hospital of Jilin University
Locations (1):
- The First Affiliated Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No